CLINICAL TRIAL: NCT06023979
Title: Early Protected Full Weight-bearing vs. Partial Weight-bearing After Surgical Fixation of Unstable Ankle Fractures, Monitored With Bio-feedback Insoles. A Single Blinded Randomized Controlled Study
Brief Title: Early Protected Full Weight-bearing vs. Partial Weight-bearing After Surgical Fixation of Unstable Ankle Fractures, Monitored With Bio-feedback Insoles.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Primoz Potocnik, Dr. med. Primoz Potocnik, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC Nr. 2023-01242
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Post Operative Treatment After Unstable Malleolar Fractures
Keywords: malleolar fractures; postoperative treatment protocol; full weight bearing; partial weight bearing; bio-feedback insoles
MeSH Terms: interventions — Partial Weight-Bearing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full weight bearing (Experimental): After 2 weeks after surgery the arm will begin full weight bearing
  Interventions: Other: Full weight bearing
- Partial weight bearing (Active Comparator): The arm will perform partial weight bearing for 6 weeks after surgery
  Interventions: Other: Partial weight bearing

INTERVENTIONS:
Other: Full weight bearing — Full weight bearing monitored with a bio-feedback insole
  Arms: Full weight bearing
Other: Partial weight bearing — Partial weight bearing monitored with a bio-feedback insole
  Arms: Partial weight bearing

SUMMARY:
The purpose of this study is to compare the postoperative results after ORIF (Open Reduction Inner Fixation) with a partial weight-bearing protocol versus an early full weight-bearing protocol. But in addition, we will measure every patient's actual load by the means of walker integrated bio-feedback insoles for the first six postoperative weeks to record the adherence to the protocol.

DETAILED DESCRIPTION:
This study aims to compare the postoperative results after PWB (partial weight bearing) and early FWB (full weight bearing) and to show, that documented early protected weight-bearing after surgical fixation of unstable ankle fractures leads to an improved early clinical outcome and a faster return to work compared to PWB. It also aims to show, that an early FWB is safe in terms of complication rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with surgically stabilized unstable ankle fractures
* signed informed consent
* closed tibial and fibular epiphysis
* age 18 or older

Exclusion Criteria:

* dementia and other known cognitive impairment or incapacity of judgement
* polytrauma
* bilateral injury of the lower extremities
* additional injury of the ipsilateral lower extremity which prevents full weight bearing
* associated injury of one or both upper extremities
* open fractures grade II° and III°
* chronic loss of sensation on plantar aspect of the feet due to known distal neuropathy
* open epiphysis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Manchester Oxford Foot and Ankle Questionnaire | 1 year
  Patient reported Outcome measure

SECONDARY OUTCOMES:
other PROMs (patient reported outcome measures) | 1 year
Range of Motion | 1 year
Secondary dislocation of fracture | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Canton Hospital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No